CLINICAL TRIAL: NCT06336356
Title: A Randomised, Double-blind, Placebo-controlled Study to Evaluate Cortisol Reserve in Response to Adrenocorticotropic Hormone Stimulation Test Following Treatment With Baxdrostat for 8 Weeks in Participants With Uncontrolled Hypertension
Brief Title: A Study to Evaluate Cortisol Reserve in Response to Adrenocorticotropic Hormone (ACTH) Stimulation Test Following Baxdrostat Treatment Compared to Placebo in Participants With Uncontrolled Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6970C00011
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Uncontrolled Hypertension
Keywords: Adrenocorticotropic hormone stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Baxdrostat 2 mg (Experimental): Participants will receive baxdrostat 2 mg tablet orally once daily.
  Interventions: Drug: Baxdrostat
- Arm 2: Placebo (Placebo Comparator): Participants will receive placebo tablet orally once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baxdrostat — Baxdrostat will be administered orally once daily.
  Other Names: RO6836191,; CIN-107
  Arms: Arm 1: Baxdrostat 2 mg
Drug: Placebo — Placebo will be administered orally once daily.
  Arms: Arm 2: Placebo

SUMMARY:
The main purpose of this study is to assess the serum free cortisol response after ACTH stimulation test at baseline and at Week 8 in participants with uncontrolled hypertension.

DETAILED DESCRIPTION:
This is a placebo-controlled study to evaluate cortisol reserve after ACTH stimulation test following treatment with 2 milligrams (mg) baxdrostat versus placebo.

The study consists of 3 period:

* 4-week screening period.
* An 8-week double-blind treatment period.
* A safety follow-up 2 weeks after last dose.

Participants will be randomized in a 2:1 ratio to one of 2 treatment arms:

1. Baxdrostat
2. Placebo

Participants will receive either baxdrostat or placebo.

The overall study duration will be up to 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants with mean seated systolic blood pressure (SBP) on automated office blood pressure measurement (AOBPM) greater than equal to (>=) 130 millimeter of mercury (mmHg) and less than (<) 170 mmHg at screening.
* Participants with mean seated SBP on AOBPM of >=130 mmHg and < 170 mmHg at randomization.
* Participants must have a stable regimen of >=1 antihypertensive medication (at least one should be a diuretic), for at least 4 weeks prior to screening.
* Participants must have an estimated glomerular filtration rate (eGFR) >=45 milliliter per minute (mL/min)/1.73-meter square (m^²) at screening.
* Participants must have a serum potassium+ (K+) level >=3.5 and < 5.0 millimole per liter (mmol/L) at screening.

Exclusion Criteria:

* Mean seated diastolic blood pressure (DBP) on AOBPM >=110 mmHg at randomization.
* Prior treatment (within the 4 weeks before screening) with angiotensin receptor Blocker (ARBs) and angiotensin converting enzyme inhibitor (ACEIs) (both taken simultaneously).
* Serum sodium (Na+) level < 135 millimole per liter (mmol/L) at screening, determined as per central laboratory.
* New York heart association functional heart failure (HF) Class IV at screening.
* Planned percutaneous coronary intervention/coronary artery bypass grafting or percutaneous coronary intervention/coronary artery bypass grafting done within 6 months prior to screening.
* Uncontrolled diabetes with glycated haemoglobin (HbA1c) > 10.0% (86 mmol/mol) at screening.
* Fridericia's corrected QT (QTcF) value > 470 milliseconds (ms) at screening, unless having a pacemaker.
* Heart rate < 45 or > 110 beats/min in a resting position, as per vital signs assessment.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Research Site, Phoenix, Arizona
  - Research Site, Tempe, Arizona
  - Research Site, Montclair, California
  - Research Site, Tarzana, California
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Metairie, Louisiana
  - Research Site, Houston, Texas
  - Research Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via there quest portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6970C00011&attachmentIdentifier=bdbb74fb-8ef9-4b33-83b5-5bf4cb03c188&fileName=CSP_D6970C00011_Redacted.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6970C00011&attachmentIdentifier=eba7230d-06f3-45ba-86d4-98134806548e&fileName=Statistical_Analysis_Plan_D6970C00011_Redacted.pdf&versionIdentifier=
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6970C00011&attachmentIdentifier=da008a0d-587f-4eb9-ba40-fff9c5607c8b&fileName=CSR_Synopsis_D6970C00011_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 10 sites in the United States of America from 10-June-2024 to 04-Dec-2024. The analyses presented in this report are based on a clinical data cutoff date of 28 January 2025.
Pre-assignment Details: Participants who met all the inclusion and none of the exclusion criteria were enrolled in this study. All study assessments were performed as per the schedule of assessment.
Groups:
- Baxdrostat 2 mg: Participants received a baxdrostat 2 mg tablet orally once daily.
- Placebo: Participants received placebo as a tablet orally once daily.
Period: Overall Study
Arm/Group | Baxdrostat 2 mg | Placebo
Started | 32 | 16
Completed | 30 | 16
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow Up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants who received at least one dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Baxdrostat 2 mg | Placebo | Total
Number analyzed (Participants) | 32 | 16 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (9.2) | 66.1 (7.4) | 64.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 26
  Male | 15 | 7 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 12 | 7 | 19
  White | 20 | 9 | 29

OUTCOME MEASURES:

1. Secondary Outcome: Incidence of Abnormal Stimulated Cortisol at Week 8
Description: The secondary endpoint is the incidence of abnormal stimulated cortisol after ACTH stimulation test at Week 8. Incidence of normal stimulated serum total cortisol level at baseline are presented.
  Normal cortisol levels are defined as at least 18 μg/dL when measured 60 minutes (±10 minutes) after stimulation. If the Week 8 results show abnormal levels, a repeat test is conducted. In this repeat test, cortisol is considered abnormal only if both of the following conditions are met: the level is less than 14.8 μg/dL at 30 minutes (± 5 minutes) and less than 18 μg/dL at 60 minutes (±10 minutes). Participants who had abnormal cortisol levels at the start of the study (baseline) were not included in this analysis.
Time Frame: Week 8
Population: The full analysis set included all randomized participants who received at least one dose of study intervention. Here, 'number of participants analyzed' and 'number analyzed' specifies participants evaluated for this outcome measure at specific timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Baxdrostat 2 mg | Placebo
Number analyzed (Participants) | 26 | 15
Participants
  Abnormal Stimulated cortisol at Week 8 | 0 | 0
  Normal Stimulated cortisol at Week 8 | 26 | 15

2. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Adverse Events of Special Interest (AESIs)
Description: Safety and tolerability of baxdrostat as compared with placebo was assessed. For this clinical study, AESIs include the following: hyperkalaemia, hyponatraemia and hypotension events that require medical intervention.
Time Frame: From Day 1 up to Week 8 or Safety follow-up (14 days post last dose), which ever comes first (up to 10 weeks)
Population: The full analysis set included all randomized participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Baxdrostat 2 mg | Placebo
Number analyzed (Participants) | 32 | 16
Participants
  Any AE | 10 | 6
  Any SAE | 0 | 0
  Any SAE with outcome death | 0 | 0
  Any AE leading to discontinuation of IP | 1 | 0
  Any possibly related AE | 6 | 3
  Any possibly related SAE | 0 | 0
  Any AESIs | 1 | 0

3. Primary Outcome: Number of Participants With Serum Total Cortisol Level Before and After Adrenocorticotropic Hormone (ACTH) Stimulation Test
Description: The primary endpoint is individual participant's cortisol levels at each timepoint. Number of participants with normal stimulated serum total cortisol level at baseline are presented here.
  Characterisation of the serum total cortisol levels before and after ACTH stimulation test. An ACTH stimulation test using 250 μg ACTH was performed at baseline and Week 8 (End of Treatment), with serum cortisol level measured before and after ACTH stimulation test.
  Normal cortisol levels are defined as at least 18 μg/dL when measured 60 minutes (±10 minutes) after stimulation. If the Week 8 results show abnormal levels, a repeat test is conducted. In this repeat test, cortisol is considered abnormal only if both of the following conditions are met: the level is less than 14.8 μg/dL at 30 minutes (± 5 minutes) and less than 18 μg/dL at 60 minutes (±10 minutes).
Time Frame: Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Baxdrostat 2 mg | Placebo
Number analyzed (Participants) | 26 | 15
Participants
  Abnormal Stimulated cortisol at Week 8 | 0 | 0
  Normal Stimulated cortisol at Week 8 | 26 | 15

ADVERSE EVENTS:
Time Frame: From Day 1 up to Week 8 or Safety follow-up (14 days post last dose), which ever comes first (up to 10 weeks)
Arm/Group | Baxdrostat 2 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/16
Other Adverse Events (participants affected / at risk) | 6/32 | 6/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baxdrostat 2 mg (N=32) | Placebo (N=16)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information may be disclosed without prior written approval from AstraZeneca.

DOCUMENTS (2):
  • Study Protocol (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT06336356/Prot_002.pdf
  • Statistical Analysis Plan (2024-12-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT06336356/SAP_003.pdf